CLINICAL TRIAL: NCT01446874
Title: Prevention of Postoperative Pneumonia (POPP Study): A Study to Evaluate the Use of a Prophylactic Clinical Strategy to Prevent Postoperative Pneumonia in Patients Undergoing Thoracic Surgery
Brief Title: Prevention of Post-operative Pneumonia (POPP)
Acronym: POPP
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Slow patient accrual and plans to perform multi-center study
Sponsor: Washington University School of Medicine (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 201106336
Record Dates: First submitted 2011-09-30; First posted 2011-10-05 (Estimated); Results first posted 2018-06-12 (Actual); Last update posted 2018-11-08 (Actual); Status verified 2018-10

CONDITIONS: Post-operative Pneumonia; Lung Cancer; Esophageal Cancer
Keywords: Incidence of post-operative pneumonia in patients undergoing surgery for primary lung cancer or primary esophageal cancer
MeSH Terms: conditions — Lung Neoplasms; Esophageal Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Pre-operative brushing (Pilot Portion) (Experimental): -Toothbrushing 3 times/day for at least 5 days preoperatively using a 0.12% chlorhexidine solution
  Interventions: Drug: 0.12% chlorhexidine solution
- Pre-operative & Post-Operative Brushing (Esophageal Resection) (Experimental): * Toothbrushing 3 times/day for at least 5 days preoperatively using a 0.12% chlorhexidine solution
  * The intensive toothbrushing regimen and chlorhexidine mouthwash will be continued for the duration of the hospitalization or a minimum of 5 days postoperatively in the study group.
  Interventions: Drug: 0.12% chlorhexidine solution
- Pre-operative & Post-Operative Brushing (Lung Resection) (Experimental): * Toothbrushing 3 times/day for at least 5 days preoperatively using a 0.12% chlorhexidine solution
  * The intensive toothbrushing regimen and chlorhexidine mouthwash will be continued for the duration of the hospitalization or a minimum of 5 days postoperatively in the study group.
  Interventions: Drug: 0.12% chlorhexidine solution

INTERVENTIONS:
Drug: 0.12% chlorhexidine solution — Toothbrushing 3 times/day for at least 5 days preoperatively using a 0.12% chlorhexidine solution and for the duration of the hospitalization or 5 days postoperatively.

SUMMARY:
Postoperative pneumonia is a major complication in patients undergoing thoracic surgery. It leads to considerable morbidity and contributes to perioperative morbidity. There is evidence in literature that supports the use of strategies for improved oral hygiene and specialized endotracheal tubes in preventing ventilator associated pneumonia (VAP) in mechanically ventilated patients. This study aims at utilizing a combination of these interventions in the perioperative period in patients undergoing planned thoracic surgical procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with lung lesions undergoing anatomic resection (lobectomy/segmentectomy/bilobectomy/pulmonary sleeve resection/pneumonectomy)
2. Patients with poor lung function (FEV1% <50% or DLCO<50% predicted or home oxygen requirement) and lung lesions undergoing non-anatomic lung resection (i.e. wedge resection).
3. Patients undergoing esophageal resection.

Exclusion Criteria:

1. Patients with ongoing symptomatic dental infections.
2. Patients with recent/ongoing pneumonia (<15 days from initial surgical patient evaluation).
3. Patients who've received a therapeutic course of antibiotics within 15 days prior to thoracic surgery.
4. Patients with a preexisting tracheostomy.
5. Age<18
6. Patients with an allergy to Peridex/chlorhexidine solution

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2011-09-22 (Actual); Primary Completion 2015-12-13 (Actual); Study Completion 2015-12-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Varun Puri, M.D., Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Semenkovich TR, Frederiksen C, Hudson JL, Subramanian M, Kollef MH, Patterson GA, Kreisel D, Meyers BF, Kozower BD, Puri V. Postoperative Pneumonia Prevention in Pulmonary Resections: A Feasibility Pilot Study. Ann Thorac Surg. 2019 Jan;107(1):262-270. doi: 10.1016/j.athoracsur.2018.08.008. Epub 2018 Oct 3. PMID 30291834
- See also: Alvin J. Siteman Cancer Center at Barnes-Jewish Hospital and Washington University School of Medicine — http://www.siteman.wustl.edu

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study opened to participant enrollment on 09/22/2011 and closed to participant enrollment on 06/08/2016.
Groups:
- Pre & Post Operative Brushing (Esophageal Resection); Pre & Post Operative Brushing (Lung Resection): * Toothbrushing 3 times/day for at least 5 days preoperatively using a 0.12% chlorhexidine solution
  * The intensive toothbrushing regimen and chlorhexidine mouthwash will be continued for the duration of the hospitalization or a minimum of 5 days postoperatively in the study group.
Period: Overall Study
Arm/Group | Pre-operative Brushing (Pilot Portion) | Pre & Post Operative Brushing (Esophageal Resection) | Pre & Post Operative Brushing (Lung Resection)
Started | 20 | 50 | 80
Completed | 18 | 46 | 62
Not Completed | 2 | 4 | 18
Not completed — Not eligible | 1 | 0 | 0
Not completed — No surgery/No qualifying surgery | 1 | 0 | 12
Not completed — Non-compliance | 0 | 4 | 0
Not completed — Antibiotics for pre-op infection | 0 | 0 | 2
Not completed — Withdrawal by Subject | 0 | 0 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pre-operative Brushing (Pilot Portion) | Pre-operative & Post-Operative Brushing (Esophageal Resection) | Pre-operative & Post-Operative Brushing (Lung Resection) | Total
Number analyzed (Participants) | 20 | 50 | 62 | 132
Age, Continuous [Median (Full Range); unit: years] | 66 [42 to 83] | 58 [24 to 77] | 63 [47 to 88] | 62 [24 to 88]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 9 | 29 | 45
  Male | 13 | 41 | 33 | 87
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 20 | 50 | 62 | 132

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Develop Postoperative Pneumonia in the Two Groups: Lung Cancer Resection Patients and Esophageal Resection Patients
Description: Patients will be considered to have postoperative pneumonia if they meet three of the following criteria within 30 days after surgery;
  1. Fever (Temperature >38.2 C)
  2. Leucocytosis (WBC>12,000/cu mm)
  3. New infiltrate on chest X-ray
  4. Positive sputum or bronchial culture
  5. Treatment with antibiotics These criteria are utilized by the national Society of Thoracic Surgeons' database.
Time Frame: Within 30 days of surgery
Population: -None of the participants from the pilot portion are included in this outcome measure as the pilot portion only measured compliance of pre-operative toothbrushing.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Brushing (Pilot Portion) | Pre-operative & Post-Operative Brushing (Esophageal Resection) | Pre-operative & Post-Operative Brushing (Lung Resection)
Number analyzed (Participants) | 0 | 46 | 62
Participants |  | 5 | 1

2. Primary Outcome: Adherence to the Pre-operative Toothbrushing Regimen
Time Frame: Completion of pre-operative toothbrushing (three times a day for 5 days prior to surgery)
Population: This outcome measure was for only the pilot portion of the study.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Brushing (Pilot Portion) | Pre-operative & Post-Operative Brushing (Esophageal Resection) | Pre-operative & Post-Operative Brushing (Lung Resection)
Number analyzed (Participants) | 18 | 0 | 0
Participants | 16 |  |

3. Secondary Outcome: Compliance With Oral Hygiene Regimen as Measured by a Daily Brushing Diary
Time Frame: Within 30 days of surgery (comparing pre-op and post-op)
Population: The Pilot Portion is not included in this outcome measure. 3 participants in the esophageal resection group was not evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Brushing (Pilot Portion) | Pre-operative & Post-Operative Brushing (Esophageal Resection) | Pre-operative & Post-Operative Brushing (Lung Resection)
Number analyzed (Participants) | 0 | 43 | 62
Participants
  Pre-op (compliant ≥ 80% of the time) |  | 39 | 50
  Pre-op (compliant 60-79.9% of the time) |  | 4 | 9
  Pre-op (compliant 40-59.9% of the time) |  | 0 | 1
  Pre-op (compliant ≤39.9% of the time) |  | 0 | 2
  Post-op (compliant ≥ 80% of the time) |  | 26 | 28
  Post-op (compliant 60-79.9% of the time) |  | 3 | 7
  Post-op (compliant 40-59.9% of the time) |  | 6 | 5
  Post-op (compliant ≤39.9% of the time) |  | 8 | 22

4. Secondary Outcome: Compliance With Oral Hygiene Regimen as Measured by the Number of Participants Who Completed the Modified Morisky Medication/Intervention Adherence Scale and Knowledge Questionnaire
Description: Compliance is measured by the number of participants who completed the Modified Morisky Medication/Intervention Adherence Scale and Knowledge Questionnaire
Time Frame: Within 30 days of surgery
Population: None of the participants from the pilot portion are included in this outcome measure as the pilot portion only measured compliance of pre-operative toothbrushing and the participants did not complete the questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Brushing (Pilot Portion) | Pre-operative & Post-Operative Brushing (Esophageal Resection) | Pre-operative & Post-Operative Brushing (Lung Resection)
Number analyzed (Participants) | 0 | 46 | 62
Participants |  | 46 | 62

5. Secondary Outcome: Perioperative Mortality
Time Frame: Within 30 days of surgery
Population: None of the participants from the pilot portion are included in this outcome measure as the pilot portion only measured compliance of pre-operative toothbrushing.
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Brushing (Pilot Portion) | Pre-operative & Post-Operative Brushing (Esophageal Resection) | Pre-operative & Post-Operative Brushing (Lung Resection)
Number analyzed (Participants) | 0 | 46 | 62
Participants |  | 0 | 3

6. Secondary Outcome: Postoperative Respiratory Failure
Description: Postoperative respiratory failure = need for postoperative mechanical ventilation, need for bronchoscopy for atelectasis, need for tracheostomy
Time Frame: Within 30 days of surgery
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Brushing (Pilot Portion) | Pre-operative & Post-Operative Brushing (Esophageal Resection) | Pre-operative & Post-Operative Brushing (Lung Resection)
Number analyzed (Participants) | 0 | 46 | 62
Participants
  Bronchoscopy for atelectasis |  | 1 | 1
  Trachestomy |  | 1 | 1
  Respiratory failure |  | 5 | 5
  Reintubation |  | 4 | 0

7. Secondary Outcome: Incidence of Fever
Time Frame: Within 24 hours of surgery
Population: as for outcome 5
Measure: Count of Participants; unit: Participants
Arm/Group | Pre-operative Brushing (Pilot Portion) | Pre-operative & Post-Operative Brushing (Esophageal Resection) | Pre-operative & Post-Operative Brushing (Lung Resection)
Number analyzed (Participants) | 0 | 46 | 62
Participants |  | 7 | 0

ADVERSE EVENTS:
Arm/Group | Pre-operative Brushing (Pilot Portion) | Pre-operative & Post-Operative Brushing (Esophageal Resection) | Pre-operative & Post-Operative Brushing (Lung Resection)
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/50 | 0/62
Other Adverse Events (participants affected / at risk) | 0/20 | 0/50 | 1/62
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pre-operative Brushing (Pilot Portion) (N=20) | Pre-operative & Post-Operative Brushing (Esophageal Resection) (N=50) | Pre-operative & Post-Operative Brushing (Lung Resection) (N=62)
Allergic reaction (Immune system disorders) | 0 | 0 | 1

LIMITATIONS AND CAVEATS:
Please note that the data for this study was reanalyzed prior to submitting manuscript and the analysis showed some of the results submitted previously to clinicaltrials.gov was incorrect. The data has now been corrected in clinincaltrials.gov.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes